CLINICAL TRIAL: NCT00235664
Title: Prospective Study of Drug Resistant Pathogens Among Liver, Intestinal and Multivisceral Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: David Paterson, MD, UPMC
Other Study IDs: IRB# 0504102
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Transplantation
Keywords: liver transplant recipients; intestinal transplant recipients; multivisceral transplant recipients

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.

INTERVENTIONS:
Procedure: Collection of stool and endotracheal aspirate samples — collection of samples

SUMMARY:
Infections caused by multidrug resistant bacteria have become more prevalent at many tertiary care and academic centers. These infections are associated with increased morbidity and mortality. The initial empiric antibiotic choice may not be adequate and delay in initiating appropriate therapy is a reason for poorer outcomes. Furthermore, not uncommonly the only therapeutic options available are associated with significant toxicity. This is a particular challenge for solid organ transplant recipients, who are immunosuppressed and have a higher risk of acquiring infections. Exposure to different classes of antibiotics has been linked to development of antibiotic resistance. Determining the risk factors for acquisition of drug-resistant bacteria and the molecular mechanisms by which resistance occurs would allow the development and implementation of strategies to minimize these infections and therefore improve outcomes. We, the researchers at the University of Pittsburgh, aim to collect surveillance cultures on patients undergoing liver, intestinal and multivisceral transplantation in order to determine the prevalence and risk factors for Pseudomonas aeruginosa (P. aeruginosa), extended-spectrum β-lactamases (ESBL)-Klebsiella and methicillin-resistant Staphylococcus aureus (MRSA), as well as determine the molecular mechanisms associated with the development of resistance in P. aeruginosa.

DETAILED DESCRIPTION:
Methods:

Day 1 is when patients are admitted to the Transplant intensive care unit (ICU) following liver, intestinal or multivisceral transplantation. Stool samples (in the case of patients with rectal bags and/or diarrhea) for cefotaxime-resistant Gram negative rods would be obtained within 24 hours of admission to the ICU and weekly thereafter until discharge from the hospital or isolation of MDR P. aeruginosa and ESBL- K. pneumoniae, whichever occurs first. While patients are intubated, endotracheal aspirates would also be obtained on a weekly basis. Nasal swabs for MRSA would be obtained within 24 hours of admission to the ICU and weekly thereafter until discharge from the hospital or isolation of MRSA, whichever comes first.

If there are no bowel movements on the days that stool is to be collected, a rectal swab will be obtained. In addition, if the endotracheal tube is pulled, no further endotracheal aspirates will be obtained. Samples will only be obtained if available. If the swab obtained on day 1 is positive for the organisms being studied, no further samples will be obtained.

No pregnancy testing will occur since all potential patients undergoing transplant must not be pregnant. Pregnant women, or women who are currently breast-feeding an infant, will not be allowed to take part in this study.

Once a drug-resistant organism (MDR P. aeruginosa, ESBL K. pneumoniae and/or MRSA) is isolated, skin swabs from the groin and subclavian areas will be obtained once. No further swabs will be obtained from the patient but he/she will be followed clinically to determine the impact of the organism on the patient's clinical outcome.

Cultures obtained at the discretion of the treating physician will be reviewed and if P. aeruginosa, ESBL-K. pneumoniae or MRSA are isolated, they will be collected from the diagnostic microbiology laboratory and stored in Dr. Paterson's laboratory for further analysis of molecular mechanisms of resistance. These samples would have been discarded once identification and susceptibility testing is completed by the diagnostic lab.

The following information will also be collected: demographic data (address, date of birth, etc.) which includes age, sex, height, weight, and state of birth, previous reports associated with the participant's condition, laboratory results, current medication use, and any other prior medical problems/history, history of prior admission, reason for transplantation, history of prior transplantation, immunosuppression used, antimicrobials received, other surgeries performed, duration of mechanical ventilation, requirement for dialysis, microbiological studies available, simplified acute physiologic score (SAPS) on admission, duration of ICU stay. This information will be obtained from the medical records and/or the subject and become part of the research record.

The patient will be seen as an inpatient at the University of Pittsburgh Medical Center and each visit will take approximately 30 minutes. The patient will be seen by a member of the research team.

Sample storage of the organism

The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. All samples will be provided de-identified. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in Dr Paterson's laboratory in Scaife Hall, Room 812, 3550 Terrace Street, Pittsburgh, PA.

The patient has completed the study once the patient is discharged from the hospital.

Laboratory methods:

Swabs for P. aeruginosa and ESBL-K. pneumoniae will be planted on cetrimide agar and nutrient agar supplemented with cefotaxime, vancomycin and amphotericin B. Antimicrobial susceptibility testing will be performed using disk diffusion test and E-test. ESBL screening will be performed using double disk diffusion test and E-test with cefotaxime-cefotaxime/clavulanic acid and ceftazidime-ceftazidime/clavulanic acid.

Swabs for MRSA will be planted in a chromogenic media selective for MRSA.

In order to study the molecular mechanisms responsible for the development of antimicrobial resistance among the P. aeruginosa isolates, quantitative real-time PCR on genes encoding common efflux pumps, PCR for mutations in quinolone resistance determining regions gyrA, gyrB and parC genes and PCR for beta-lactamases will be performed.

Pulsed-field gel electrophoresis (PFGE) will be performed on the isolates of each single patient, to determine if the isolates are genotypically similar. PFGE will also be done in all MDR P. aeruginosa isolates in order to determine if they belong to a single or multiple clones within the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU who are identified as having undergone liver, intestinal or multivisceral transplantation. This includes cadaveric and living related liver transplants.
* Patients must be above 18 years of age.
* Patients undergoing re-transplantation may also be included.
* Written informed consent from patient or a proxy.

Exclusion Criteria:

* Known colonization or infection with multidrug resistant (MDR) P. aeruginosa, MRSA or ESBL-Klebsiella prior to admission to the ICU.
* Pregnancy or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in ICU who are identified as having undergone liver, intestinal or multivisceral transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-10; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States